CLINICAL TRIAL: NCT06937944
Title: A Phase 3 Clinical Study to Evaluate the Efficacy and Safety of Recombinant Botulinum Toxin Type A for Injection (Eveotox) Compared With a Single Treatment of Botox and Placebo,and Repeated Treatment of Eveotox in Moderate to Severe Glabellar Lines
Brief Title: Efficacy and Safety of Recombinant Botulinum Toxin Type A (Eveotox) for Injection to Treat Moderate to Severe Glabellar Lines
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: JHM BioPharma (Tonghua) Co. , Ltd. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JHM03-CT301
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Moderate to Severe Glabellar Lines
Keywords: Moderate to Severe Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Biological: Rcombinant botulinum toxin type A for injection (Eveotox) Biological: OnabotulinumtoxinA (Botox) Biological: : Placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eveotox (Experimental): Eveotox, 20 Units, divided into five injections into the glabellar area. Administered in double-blind fashion at cycle 1 followed by up to 3 open-label cycles.
  Interventions: Biological: Rcombinant botulinum toxin type A for injection（Eveotox)
- OnabotulinumtoxinA (Botox ) (Active Comparator): Botox,20 Units, will be administered in double-blind fashion during treatment cycle 1 only, followed by up to 3 of Eveotox(20 Units).
  Interventions: Biological: OnabotulinumtoxinA (Botox)
- Placebo (Placebo Comparator): Placebo, will be administered in double-blind fashion during treatment cycle 1 only, followed by up to 3 of Eveotox(20 Units)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rcombinant botulinum toxin type A for injection（Eveotox) — Rcombinant botulinum toxin type A for injection（Eveotox)
  Arms: Eveotox
Biological: OnabotulinumtoxinA (Botox) — OnabotulinumtoxinA (Botox)
  Arms: OnabotulinumtoxinA (Botox )
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 3 clinical study to evaluate the efficacy, safety, and immunogenicity of single/repeated injections of Eveotox in the treatment of moderate to severe glabellar lines. The study consists of Study Part 1 (randomized double-blind controlled study) and Part 2 (open-label study). Part I is a multicenter, randomized, double-blind, single-injection, active-controlled and placebo-controlled study to evaluate the efficacy, safety, and immunogenicity of Eveotox in the treatment of moderate to severe glabellar lines; Part 2 is an open-label study to evaluate the efficacy, safety, and immunogenicity of repeated injections of Eveotox in the treatment of moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are between 18 to 65 years of age
* Moderate or severe glabellar lines during maximum frown based on the Investigator Global Assessment Frown Wrinkle Severity scale
* Moderate or severe glabellar lines during maximum frown based on the Patient Frown Wrinkle Severity scale
* Willing and able to follow all trial procedures, attend all scheduled visits, and successfully complete the trial

Exclusion Criteria:

* Subjects who have a history of oversensitivity to the Botulinum Toxin A type or other components of the study drug
* Subjects who have implanted any permanent materials in the glabellar area or received semi-permanent fillers within the first 2 years of screening
* Subjects with active skin infections at the injection site or systemic skin disease, which the investigator judges can affect the evaluation of efficacy or safety
* Subjects who have a history of injecting drugs similar to the study drug within 6 months prior to selection or are foreseen to use during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | Within 4 weeks
  Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement of ≥ 2 points in FWS score (at maximum frown) at week 4 visit relative to baseline, based on both the investigators´ and the subjects´ in-clinic assessments.

SECONDARY OUTCOMES:
Secondary Outcome Measure | Within 52 weeks
  Incidence of serious adverse events and drug-related adverse events during the study.

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Xianyang Hospital of Yan'an University, Xianyang, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Affiliated Hangzhou First People's Hospital, School of Medicine, Westlake University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No